CLINICAL TRIAL: NCT02791750
Title: 5 Years Follow-up in the Lorraine Institute of Oncology With Adjuvant Therapy for Women With Breast Invasive Carcinoma
Brief Title: 5 Years Follow-up With Adjuvant Therapy for Women With Breast Invasive Carcinoma
Acronym: HACAMI
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL OBS 02
Record Dates: First submitted 2016-05-25; First posted 2016-06-07 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: hormone replacement therapy; breast cancer; follow up
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Patients followed for a medical consultation in the Institut de Cancérologie de Lorraine at 5 years of the beginning of an adjuvant hormonal therapy.
  Interventions: Other: questionnary of quality of life

INTERVENTIONS:
Other: questionnary of quality of life

SUMMARY:
Non-persistence to adjuvant hormonal therapy for breast cancer at 5 years decrease its efficacy. The objective of this study is to know the women experience (persistence, treatment changes, quality of life) and its determinants, in a french population.

ELIGIBILITY:
Inclusion Criteria:

* Patients following-up in the Lorraine Institute of Oncology at 5 years of the beginning of an adjuvant hormonal therapy
* Women with breast invasive carcinoma positive-RH and indication of adjuvant hormonal therapy
* Adult patients
* Being capable and agree to follow the study procedure
* Patients informed and non-opposed
* Covered by social security

Exclusion Criteria:

* History of other cancer except basal cell carcinoma
* Patients with breast invasive carcinoma negative-RH
* Synchronous metastases
* Relapsed
* Previous adjuvant hormonal therapy
* Men
* Patients with guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients following-up in the Lorraine Institute of Oncology at 5 years of the beginning of an adjuvant hormonal therapy
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-03 (Actual)

PRIMARY OUTCOMES:
Factors associated with persistence to hormone therapy for breast cancer | 1 day
  Women will be classed as persistent if they don't discontinue or abandon hormone therapy during the 5 years after the introduction of the medication. The information will be recorded thanks to a self-questionnary fulfilled the inclusion day.
  The baseline characteristics will be compared between persistent women and non-persistent women.

SECONDARY OUTCOMES:
Comparison of the quality of life | 1 day
  Quality of life between patients who continued hormone therapy for 5 years and patients who discontinued treatment early will be searched for using the questionnaire
Proportion of women with a change in their treatment | 1 day
  Proportion of women who have changed treatment within 5 years following the placing on hormone therapy and reasons for the change.
Cause of treatment discontinuation | 1 day
  In the subgroup of women who stopped hormone therapy within 5 years following the hormone therapy, determination of the treatment discontinuation.
Continued homonotherapy | 1 day
  In the subgroup of women who have been treated with hormone therapy for 5 years, determine the proportion of women not opposed to the continuation of hormone therapy beyond 5 years

CONTACTS AND LOCATIONS:
Overall Officials: LESUR ANNE, Md, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No